CLINICAL TRIAL: NCT06838689
Title: Participatory Approach to Qualitative Research (PAQ): Comparing Two Methods of Engaging Stakeholders in Qualitative Research
Brief Title: Participatory Approaches to Qualitative Research (PAQ): Comparing Two Approaches to Patient, Public and Clinician Involvement in Qualitative Research
Acronym: PAQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Catherine Hylas Saunders, Assistant Professor of Medicine and of Health Policy and Clinical Practice, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PAQ_STUDY02002675_RCT; SOE-2023C3-25572 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2025-02-19; First posted 2025-02-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Mental Health Services; Cancer Screening; Serious Illness
Keywords: Pediatric mental health; Serious illness in elderly patients; cancer screening

STUDY DESIGN:
Intervention Model Description: Experimental Intervention 1: Consultative PPCI Model via Community Advisory Boards (CAB): Community Advisory Board: a consultative model of engagement where participants attend 4 quarterly meetings with shared leadership between participants and research team.
  Experimental Intervention 2: Collaborative PPCI Model via the Participatory Approach to Qualitative Research (PAQ) Participatory Approach to Qualitative Research: a collaborative model of engagement with 4 idea coproduction sessions and a close partnership with study staff.
Who Masked: Outcomes Assessor
Masking Description: Researchers analyzing the data remain blinded to group allocation to minimize bias in data interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consultative PPCI Model via Community Advisory Boards (CAB) (Experimental): Community Advisory Board: a consultative model of engagement where participants attend 4 quarterly meetings with shared leadership between participants and research team.
  Interventions: Other: Comparison of two standard of care regimens
- Collaborative PPCI Model via the Participatory Approach to Qualitative (Experimental): Participatory Approach to Qualitative Research: a collaborative model of engagement with 4 idea coproduction sessions and a close partnership with study staff.

INTERVENTIONS:
Other: Comparison of two standard of care regimens — Participatory Approaches to Qualitative Research (PAQ): Comparing Two Approaches to Patient, Public and Clinician Involvement (PPCI) in Qualitative Research: PAQ and CAB (Community Advisory Boards)
  Other Names: Comparison between the CAB and PAQ models of community engagement
  Arms: Consultative PPCI Model via Community Advisory Boards (CAB)

SUMMARY:
The goal of this trial is to compare two types of patient, public and clinician involvement (PPCI) in research: Consultative PPCI and Collaborative PPCI.

The study team will compare these methods of PPCI in a randomized clinical trial (RCT) in which PPCI participants will engage with research teams on one of three real qualitative research interview studies addressing topics: 1) pediatric mental health, 2) cancer screening and 3) serious illness. Qualitative interviews are conversations with people about their experiences and perspectives. In all three qualitative studies, PPCI participants will help us at every stage of the research, from design (making choices about how to set up the study) through dissemination (sharing findings).

The researchers do not know about any quantitative (numbers) evidence from RCTs about how well different PPCI approaches work. As far as the study team knows, this is the first RCT of PPCI approaches. Given this gap in knowledge, the research question is: How does a Consultative PPCI approach compare to a Collaborative PPCI approach in increasing engagement and partnership trust in research, particularly among historically underrepresented groups? The researchers' best guess (hypothesis), considering the information available, is that Collaborative PPCI will increase PPCI participant engagement, trust and the patient-centeredness of research more than Consultative PPCI.

DETAILED DESCRIPTION:
This stratified randomized controlled clinical trial (RCT) is to test Consultative patient, public and clinician involvement (PPCI) in research against Collaborative PPCI in the context of three real-world qualitative research studies. Qualitative research methods can reveal insights into complex health phenomena, such as access to health services, clinician-patient communication, implementation research, and organizational culture and improvement. PPCI has also been acknowledged as indispensable in enhancing the validity, rigor and credibility of research.

The research team developed detailed guides for two approaches to PPCI throughout the lifetime of qualitative research projects, including 1) design, 2) data collection, 3) analysis and 4) dissemination. While there is a strong theoretical rationale that participatory research processes like Consultative PPCI may improve partner engagement more than consultative PPCI, evidence from experimental studies is lacking.

Given this gap, the research question is: How does a Consultative PPCI approach to involvement in research compared to a Collaborative PPCI approach in increasing engagement and partnership trust in research, particularly among historically underrepresented groups?

The study team hypothesizes Collaborative PPCI will result in higher partner-reported engagement, trust and patient-centeredness of research than Consultative PPCI.

Study Aims:

1. To compare the effectiveness of Consultative PPCI versus Collaborative PPCI on partner engagement in research (primary outcome), partnership trust (secondary outcome).
2. To use mixed methods to determine whether stakeholder engagement in research and partnership trust vary based on stakeholder characteristics.
3. To evaluate the extent to which engagement and partnership trust are mediated by engagement experience and group dynamics.

The research team will conduct a randomized controlled trial (RCT) to test the relative effectiveness of these PPCI approaches across three real-world qualitative studies. Participants will be randomly assigned to Consultative or Collaborative PPCI using a stratified approach with three embedded qualitative studies as strata. The core function of Collaborative PPCI is to test a simple, collaborative partner engagement model, while the core function of Consultative PPCI is to test the traditional consultative partner engagement model. The researchers are are operationalizing Consultative PPCI with Community Advisory Boards (CAB) and Collaborative PPCI with a new approach called the Participatory Approach to Qualitative Research (PAQ). The study team selected an RCT with stratified randomization to evaluate the research question in the context of three diverse topic areas, to maintain separate Consultative and Collaborative study groups of reasonable size within each strata (n=10 for each study's CAB or PAQ group, for a total of 60 participants), and to ultimately increase generalizability of results. Following randomization, the researchers will evaluate for balance across groups in participant age, race, ethnicity, rurality and composite socioeconomic status (comprising education and income). The objectives, interventions and outcomes will be measured at the individual participant level. The RCT will be conducted over an 18-month period. The PAQ and CAB arms will have separate professional research staff facilitators, both experienced in CAB and PAQ facilitation; these facilitators will be involved in all three project strata. Prior to study start, the research team will standardize Consultative and Collaborative PPCI training.

ELIGIBILITY:
Inclusion criteria & Exclusion criteria across three sub-specialties:

Pediatric mental health

Inclusion:

* Adults aged ≥18 years
* Can communicate in English
* Able to take part in research activities via a computer or a smartphone
* Patients, care partners, clinicians, other healthcare professionals, teachers and school staff, health policy experts, and community members
* Has lived experience or professional expertise relating to pediatric mental health

Exclusion:

* Children <18 years
* Cannot communicate in English
* Adults unable to provide verbal consent
* Prisoners
* Unable to take part in research activities via a computer or a smartphone

Generalized cancer screening

Inclusion:

* Adults aged ≥21 years
* Can communicate in English
* Able to take part in research activities via a computer or a smartphone
* Patients, care partners, clinicians, other healthcare professionals, health policy experts, and community members
* Is eligible for population-based cancer screening tests (breast, prostate, cervical, colorectal cancer), or has lived experience or professional expertise relating to generalized cancer screening

Exclusion:

* Children <18 years
* Cannot communicate in English
* Adults unable to provide verbal consent
* Prisoners
* Unable to take part in research activities via a computer or a smartphone

Serious illness experience

Inclusion:

* Adults aged ≥18 years
* Can communicate in English
* Able to take part in research activities via a computer or a smartphone
* Patients, care partners, clinicians, other healthcare professionals, health policy experts, and community members
* Has lived experience or professional expertise relating to serious illness (defined as "a health condition that carries a high risk of mortality and either negatively impacts a person's daily functioning or quality of life or excessively strains his or her caregivers."

Exclusion:

* Children <18 years
* Cannot communicate in English
* Adults unable to provide verbal consent
* Prisoners
* Unable to take part in research activities via a computer or a smartphone

Note: We will not specifically exclude pregnant women, so they may be included incidentally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient Engagement in Research scale (PEIRS-22) | 18 months
  Engagement in research, measured using the Patient Engagement in Research scale (PEIRS-22). Total score is 22-110, with higher scores reflecting greater engagement in research.

SECONDARY OUTCOMES:
Research Engagement Survey Tool (REST) | 18 months
  Partnership Trust, measured using the "build and maintain trust in the partnership" scale of the Research Engagement Survey Tool (REST). Component scores are calculated as means, with four being the best possible score.
Patient and Public Involvement in Research Assessment Survey | 18 months
  Research patient-centeredness, measured using the Patient and Public Involvement in Research Assessment Survey (PAS). Possible scores range from 0-80, with higher scores equating to higher patient-centeredness.
Person-Centeredness of Research Scale | 18 months
  Research patient centeredness, measured using the Person-Centeredness of Research Scale. Possible scores range from -14 to +14, with higher scores representing more patient-centered research.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Geisel School of Medicine at Dartmouth, Hanover, New Hampshire
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://healthcareexperiencelab.com/participatory-approaches-to-qualitative-research/